CLINICAL TRIAL: NCT04671277
Title: Oral Processing Behavior of Gluten-free and Gluten-containing Breads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Nicoletta Pelegrini, Associate Professor, University of Udine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0002491
Record Dates: First submitted 2020-11-30; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Oral Processing Behavior; Mastication; Swallowing
Keywords: food oral processing; gluten-free bread; mastication; texture; saliva; food bolus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chewing of breads (Experimental): 6 samples (2x3 full factorial design with 2 white sandwich bread types (a regular gluten-containing (GC) and a gluten-free version (GF)) and 3 spread conditions (no spread, butter and mayonnaise)) were evaluated in two sessions of 30 min each. The first session was designed for video recording and the second session for the evaluation of texture attributes and collection of food bolus.
  Bread samples were served as two stacked cylinders resembling the consumption of a sandwich (diameter: 3.5 cm, approximate total height: 2.4 cm) (Figure 1). Due to differences in bread density, the average weight of two stacked cylinders was 5.1 ± 0.2 and 5.7 ± 0.4 for GC and GF breads, respectively. Butter and mayonnaise were added to breads at approximately 12% w/w.
  Interventions: Other: Chewing of breads

INTERVENTIONS:
Other: Chewing of breads — During the video recording session, participants were asked to place the whole sample (5-6 g) in the mouth (e.g. single bite) and chew naturally until the bolus is ready for swallowing.
  During the second section, participants were asked to place the whole sample in the mouth and chew naturally. After 5 chewing cycles, participants checked all the attributes that describe the texture sensations perceived at the beginning of mastication. A list of attributes and their definitions were provided to guide the participants. Participants proceeded with chewing until the swallowing point when they again checked all the attributes that characterize the texture sensations perceived at the end of mastication. The food bolus was then spat in a container.

SUMMARY:
To attend the increasing demand for gluten-free products, new gluten-free formulations emerged in the market containing alternative ingredients to mimic the protein functionality of wheat. The replacement of wheat, however, has consequences in the sensorial properties of gluten-free products, which can compromise the acceptability of products. This study aims to investigate the oral processing behaviour of gluten-free and gluten-containing breads. Two commercial products, one gluten-free and one gluten-containing bread will be tested either without spread or with butter or mayonnaise. Spreads will be added to the breads to resemble a sandwich consumption which is a more realistic approach than that previously used. The investigators hypothesize that changes in the structure of gluten-free breads resulting from the absence of a strong gluten network can have a prominent impact on the way gluten-free bread is orally processed. The investigators also hypothesize that the addition of spreads will facilitate the oral processing of bread due to an increase in moisture content and lubrication.

The number of chews, number of swallows and eating duration will be determined through video recording of 20 subjects. The texture attributes predominantly at the beginning of mastication and at the swallowing point will be accessed using a check-all-that-apply test. Additionally, the amount of saliva incorporated during chewing will be determined from the spat out food bolus.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-59 years old
* Have good general oral health (self-reported)
* Have normal smell and taste functions (self-reported)
* Have a normal body mass index (BMI 18.5-24.9 kg/m2) (based on self-reported weight and height)
* Have no dental braces or a piercing in or around the mouth (except removable piercings)
* Have given written informed consent

Exclusion Criteria:

* Have any food allergy or intolerance for gluten
* Have mastication and/or swallowing problems caused by neurological problems, i.e. stroke, Parkinson, Alzheimer, Huntington
* Being pregnant or lactating (self-reported)
* Use medication that may affect the function of taste, smell, mastication and salivation

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Oral processing behavior | Day 1, approximately 30 min
  Participants were video recorded during bread consumption and the parameters number of chews, number of swallows and eating duration were extracted from the videos
Texture sensations perceived during chewing | Day 2, approximately 30 min
  Texture attributes were selected after 5 chewing cycles and at the moment of swallowing using the check-all-that-apply methodology

SECONDARY OUTCOMES:
Saliva content in food bolus | Day 2, approximately 30 min
  The amount of saliva that was incorporated in the food bolus during chewing

CONTACTS AND LOCATIONS:
Locations (1):
- Nicoletta Pellegrini, Udine, Select Region, Italy

DOCUMENTS (2):
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04671277/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04671277/Prot_SAP_001.pdf